CLINICAL TRIAL: NCT04249986
Title: Backpack Weight Impacts on Perceived Exertion and Heart Rate Variability
Brief Title: Backpack Weight Impacts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2019126
Record Dates: First submitted 2020-01-24; First posted 2020-01-31 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-08

CONDITIONS: Exertion; Excess

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The Borg Rating of Perceived Exertion between 17 and 19 lb BPW (Active Comparator): Participants will be randomized to both 17 and 19 pounds for the first hike and the alternate condition for the second hike. A random number generator will create 1 block that includes 10 participants in each block to ensure comparable numbers to subjects starting at different base backpack weight. Participants assignments will then be included in a sealed manila envelopes.
  Interventions: Behavioral: The Borg Rating of Perceived Exertion
- The Borg Rating of Perceived Exertion between 19 and 17 lb BPW (Active Comparator): Participants will be randomized to both 19 or 17 pounds for the first hike and the alternate condition for the second hike. A random number generator will create 1 block that includes 10 participants in each block to ensure comparable numbers to subjects starting at different base backpack weight. Participants assignments will then be included in a sealed manila envelopes.
  Interventions: Behavioral: The Borg Rating of Perceived Exertion

INTERVENTIONS:
Behavioral: The Borg Rating of Perceived Exertion — Participants who satisfy the exclusion criteria and health assessment instrument are categorized in the lowest risk group for cardiac events and does not require medical screening for mild to moderate exercise per ACSM guidelines.

SUMMARY:
Backpacking is an increasingly popular outdoor recreational activity. The base pack weight (BPW) includes gear that is not consumed or worn on the body: shelter, sleep system, weather-proofing layers and personal gear to ensure a degree of comfort and safety. As such, reducing BPW is one of the most important tasks a backpacker manages when preparing for a trip. Available recommendations for ideal BPW are currently inconsistent, lack clear parameters, and rely on anecdotal evidence. The study aims to collect field data on perceived exertion and heart rate (HR) in relation to BPW during a day-long interval of hiking. Such findings can have implications on the cost and safety profiles extending from recreational backpacking to military and wilderness rescue operations.

ELIGIBILITY:
Inclusion Criteria:

* Only adult (age 18-65)
* Have gone on at least two overnight backpacking trips in the past 5 years
* Have hiked at least 8 miles in a day on one of those trips

Exclusion Criteria:

* Lower extremity injuries or surgeries in the past 6-months
* Daily Smokers
* Chronic medical problems:
* Hypertension
* High cholesterol
* Diabetes
* Heart attack
* Heart surgery, cardiac catheterization, or coronary angioplasty
* Pacemaker/implantable cardiac defibrillator/rhythm disturbance
* Heart valve disease
* Heart failure
* Heart transplantation
* Congenital heart disease
* Kidney disease
* Back pain

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-02-21 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
The Borg Rating of Perceived Exertion During the Total Hike | 2 weeks
  Participants will report their perceived exertion towards the end of both hikes. The Borg Rating of Perceived Exertion scale ranges from 6 to 20. 6 being the lowest score of no exertion and 20 being the highest of maximal exertion.

SECONDARY OUTCOMES:
Heart Rate | 2 weeks
  Difference between participants' heart rate during both 17 and 19 pound base backpack weight.
The Borg Rating of Perceived Exertion During Incline and Decline Sections of the participant | 2 weeks
  Participants will report the perceived exertion mid-hike and towards the end. The Borg Rating of Perceived Exertion scale ranges from 6 to 20. 6 being the lowest score of no exertion and 20 being the highest of maximal exertion.

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Spano, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Fresno, Fresno, California, United States

IPD SHARING:
Plan to Share IPD: No